CLINICAL TRIAL: NCT05608655
Title: A Multicenter, Prospective, Randomized Controlled Trial to Evaluate the Efficacy and Safety of DKutting Balloon Versus Chocolate Balloon in the Treatment of Femoral and Popliteal Artery Stenosis
Brief Title: DKutting Balloon Versus Chocolate Balloon to Treat Femoral and Popliteal Artery Stenosis
Acronym: DELTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DK Medical Technology (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-P-22-005
Record Dates: First submitted 2022-10-21; First posted 2022-11-08 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Femoral Artery Stenosis; Popliteal Artery Stenosis
Keywords: PTA Scoring Balloon; Optimal Balloon Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DKutting (Experimental): DKutting LL Scoring Balloon, DK Medtech Co Ltd
  Interventions: Device: DKutting LL balloon
- Chocolate (Active Comparator): Chocolate Balloon, TriReme Medical LLC
  Interventions: Device: Chocolate balloon

INTERVENTIONS:
Device: DKutting LL balloon — After pre-dilation balloon is used (if any), DKutting LL balloon is used as final dilatation balloon before Stent implantation or Drug Coated Balloon deployment
  Arms: DKutting
Device: Chocolate balloon — After pre-dilation balloon is used (if any), Chocolate balloon is used as final dilatation balloon before Stent implantation or Drug Coated Balloon deployment
  Arms: Chocolate

SUMMARY:
A Multicenter, Prospective, Randomized Controlled Trial to Evaluate the Efficacy and Safety of DKutting Balloon Versus Chocolate Balloon in the Treatment of Femoral and Popliteal Artery Stenosis

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized controlled, open-label, noninferior study to evaluate achievement of optimal PTA dilatation. A total of 188 patients will be enrolled from 14 sites in China. All patients enrolled will be assigned to the test group (DKutting LL balloon, n=94) and the control group (Chocolate balloon, n=94) with randomized allocation ratio of 1:1.

Primary endpoint is percentage of PTA cases in which <30% diameter stenosis without a flow limiting dissection is achieved. A 30-day after procedure follow-up will be conducted for all 188 patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year-old male & non-pregnant female
* Patients with Arteriosclerosis Obliterans of Lower Extremities, including stenosis or osculation in femoropopliteal artery.
* Rutherford clinical category-Becker class: 2 to 5
* Patients understand the purpose of the study, will voluntarily participate in the study and sign informed consent. Patients are willing to undergo clinical follow-up as required by this study.
* Digital subtraction angiography (DSA) shows femoropopliteal artery stenosis above 70%, appropriate for treatment with balloon angioplasty
* Reference vessel diameter from 2.5 to 7mm; Total length of lesion is less than 200mm; Total length of osculation lesion is less than 100mm
* Only one target lesion needs to be Treated. Treatment of non-target lesion, if any, must be completed prior to treatment of target lesion and must be deemed a clinical angiographic success as visually assessed by the physician. The number non-target lesions are limited to maximum 3.

Exclusion Criteria:

* Acute or sub-acute thrombosis exist in target lesion
* Severe calcified lesion (PACSS Grading 4)
* Guidewire cannot cross target lesion
* Amputation planned within 30 days
* In-stent restenosis
* Flow-limiting dissection (NHLBI grading: D-F) occurred in target lesion by pre-dilation
* No other lumen-reduction devices (such as: cutting balloon, dual-wire balloon, Hawk, ELCA etc.) are treated before or after test/control group treatment.
* Before test/control group treatment, target lesion was expanded by Antegrade Dissection Re-entry (ADR) technique.
* Patient who cannot accept anticoagulant or antiplatelet therapy
* Aware of patient allergic to heparin, contrast, aspirin and clopidogrel, anesthetics
* Patients who have not completed clinical trials of other drugs or devices
* Patients with poor compliance and unable to complete the study, which is identified by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Achievement of Optimal PTA in Percent | 1 day
  Percentage of PTA cases in which <30% diameter stenosis without a flow limiting dissection (NHLBI grading: D-F). Residual stenosis in percent and dissection NHLBI grading are accessed by independent core-lab with Medis Suite XA based on in-procedure QCA angiography. [0-100%, higher the better]

SECONDARY OUTCOMES:
Device Success Rate in Percent | 1 day
  Device Success defined as successful delivery to the target lesion, deployment without balloon rupture, and retrieval after procedure, as qualitatively accessed by physician. [0-100%, higher the better]
Numerical Acute Lumen Gain in mm | 1 day
  In-lesion acute lumen gain defined as minimal lumen diameter (MLD) in lumen after dilatation by either arm device minus baseline MLD, as accessed by independent core-lab with Medis Suite XA based on in-procedure QCA angiography. [0-3mm, higher the better]
Technical Success Rate in percent | 0-7 days
  Percentage of target Lesion achieved <30% diameter stenosis without a flow limiting dissection (NHLBI grading: D-F) and No Adverse Event happened in hospital. [0-100%, higher the better]
Freedom from clinical-driven TLR rate in percent | 30+/-7 Days post procedure
  Freedom from clinical-driven target lesion revascularization 1 month post procedure [0-100%, higher the better]
Rutherford Grading Reduction in percent | 30+/-7 Days post procedure
  Percentage of both groups' patent number, whose Rutherford Grading [0-6, lower is reduced by at least 1 grade post procedure, compared with pre-procedure grade. [0-100%, higher the better]
Freedom from Amputation above ankle rate in percent | 30+/-7 Days post procedure
  Percentage of both groups' patient number who is free from Amputation above ankle 1 month post procedure. [0-100%, higher the better]
Numerical Ankle Brachial Index | 0-7days
  Record of both groups' patient's Ankle Brachial Index (ABI) pre/post procedure by Doppler ultrasonic stethoscope. [ABI≤0.9: confirmed peripheral artery disease; ABI≥0.97: normal people]

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Fu, Dr., Principal Investigator — Shanghai Zhongshan Hospital
Locations (14):
- China (14):
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Hospital of Chengdu Traditional Chinese Medicine University, Chengdu, Sichuan
  - The Third People's Hospital of Chengdu, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - China-Japan Friendship Hospital, Beijing
  - Xuanwu Hospital of Capital Medical University, Beijing
  - The First Affiliated Hospital of Naval Medical University, Shanghai
  - Zhongshan Hospital of Fudan University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin